CLINICAL TRIAL: NCT01459991
Title: The Mediterranean Diet and Lactation Study: A Diet Study in Lactating Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: California Walnut Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Walnut Study
Record Dates: First submitted 2011-10-24; First posted 2011-10-26 (Estimated); Last update posted 2011-10-28 (Estimated); Status verified 2011-10

CONDITIONS: Breast Feeding
Keywords: walnut; mediterranean
MeSH Terms: conditions — Breast Feeding | interventions — PR-10 protein, walnut birch pollen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mediterranean (Experimental): Participants in this arm will follow a Mediterranean style diet, rich in olive oil and fruits and vegetables, and also consume 1 ounce of walnuts daily.
  Interventions: Other: Walnut
- MyPyramid (Active Comparator)
  Interventions: Other: MyPyramid

INTERVENTIONS:
Other: Walnut — Participants will consume 1 ounce walnuts daily and follow a Mediterranean style diet.
  Arms: Mediterranean
Other: MyPyramid — Participants will follow a USDA MyPyramid style diet for lactating moms.
  Arms: MyPyramid

SUMMARY:
Purpose: During lactation, several physiological modifications occur including cellular differentiation and proliferation, as well as elevation in inflammation. The role of the Mediterranean (MED) diet rich in walnuts has been shown to favorably modify fatty acid profiles and to reduce inflammation. The study goal is to evaluate the anti-inflammatory effects of the MED diet rich in walnuts during lactation, a time of increased inflammatory response.

Procedures: A randomized, controlled dietary intervention trial among lactating women comparing the effects of a Mediterranean-style diet with walnuts to the USDA's MyPyramid Diet for Moms was commenced to determine the effects of the diet on fatty acid profiles and biomarkers of inflammation in breast milk and material serum/plasma. Secondary outcomes of interest include effects of maternal diet assignment on maternal body weight and body composition as well as infants' growth and health during the study trial period.

Population: The study population includes healthy women between the ages of 18-40 years who are within 6 months post-partum and plan to breastfeed a minimum of 3 times per day for 6 months following study entry. There have been a total of 138 participants enrolled in the study. All 138 participants are women; 34 identified themselves as Hispanic, and 104 said they were not Hispanic.

ELIGIBILITY:
Inclusion Criteria:

* plan to breastfeed 3 times daily for 6 months
* no nut allergies
* no history of cancer, renal disease, liver disease, or diabetes
* no smoking

Exclusion Criteria:

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 138 (Actual)
Dates: Start 2008-10; Primary Completion 2010-12 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Estrogen associated hormones | baseline, 2 month, 4 month, 6 month, 12 month
  To assess the effect of diet change on estrogen-associated hormones as measured by estradiol-17 beta in serum and breast milk, as well as sex hormon binding globulin (SHBG) in serum among lactating women.
inflammatory and oxidative stress biomarkers | baseline, 2, 4, 6, and 12 months
  Determine indirect/secondary effects of diet intervention on biomarkers of inflammation and oxidative stress as measured by serum high sensitivity C-reactive protein (hsCRP) and urinary 15-iso-prostaglandin-F2alpha (8-iso-PGF2alpha), respectively.
body measurements | baseline, 2, 4, 6, and 12 months
  Assess repeated measures of change in body weight and composition related to dietary group assignment.
diet adherence | Baseline, 2, 4, 6, and 12 months
  Evaluate adherence and exposure to the diet intervention using the objective plasma biomarker, alpha-linolenic acid. Alpha-linolenic acid will be measured in breast milk as well as maternal plasma as a biomarker of intake/exposure.

CONTACTS AND LOCATIONS:
Locations (1):
- Nutrition Research Clinic, Tucson, Arizona, United States